CLINICAL TRIAL: NCT05444153
Title: Efficacy and Safety of Early Initiation of Oral Semaglutide 50 mg Once Daily Versus Empagliflozin 25 mg Once Daily in Younger Patients With Newly Diagnosed Type 2 Diabetes and Obesity
Brief Title: Research Study to Compare Semaglutide Tablets With Empagliflozin Tablets Taken Once Daily in People With Type 2 Diabetes and Obesity
Acronym: PIONEER START
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4668; U1111-1270-0763 (Other: World Health Organization (WHO)); 2021-005396-39 (EudraCT Number)
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral semaglutide (Experimental): Participants will receive once daily oral semaglutide tablet for 104 weeks in a dose escalation fashion of 3milligrams (mg), 7mg, 14 mg and 25 mg once every four weeks during the first 16 weeks and a maintenance dose of 55 mg for the rest 88 weeks.
  Interventions: Drug: Semaglutide
- Empagliflozin (Active Comparator): Participants will receive once daily empagliflozin tablet for up to 104 weeks, starting with a dose of 10 mg for the first 8 weeks and the maintenance dose of 25 mg for the rest 96 weeks.
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Semaglutide — Participants will receive 1 tablet of oral semaglutide once daily.
  Arms: Oral semaglutide
Drug: Empagliflozin — Participants will receive 1 tablet of empagliflozin once daily.
  Arms: Empagliflozin

SUMMARY:
This study compares the medicines semaglutide and empagliflozin in people with newly diagnosed type 2 diabetes and obesity. The study will look mainly at how well the blood sugar and body weight are controlled when participants are taking the study medicine. Participants will either get semaglutide tablets or empagliflozin tablets. Which treatment participants get is decided by chance. Participants will get one tablet per day for 2 years. The study will last for about 2 years and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18- less than (<) 50 years at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus less than or equal to (<=) 365 days from the day of screening.
* Glycated haemoglobin (HbA1c) of 7.0-9.5 percentage (%) (53-80 millimoles per milliliter [mmol/mol]) (both inclusive).
* Body mass index (BMI) greater than or equal to (>=) 30.0 kilograms per meter square (kg/m^2).
* Treatment naïve to any antidiabetic drug(s). However, for a subset of participants (≤25%) any metformin dose or formulations administered is allowed.

Exclusion Criteria:

* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria since diagnosed with type 2 diabetes mellitus. Prior insulin treatment for gestational diabetes is allowed.
* Renal impairment measured as estimated glomerular filtration rate (eGFR) value of less than (<) 60 milliliter per minute per 1.73 meter square (1.7mL/min/1.73 m^2) at screening.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to day of screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* C-peptide less than (<)1.5 nanograms per milliliter (ng/mL) at screening.
* Positive insulinoma associated-protein 2 (IA-2) antibodies or anti-glutamic acid decarboxylase (anti-GAD) antibodies.
* History of major surgical procedures involving the stomach or small intestine potentially affecting absorption of drugs and/or nutrients.
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-06 (Estimated); Primary Completion 2024-10-02 (Estimated); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
Participants acheiving glycated haemoglobin (HbA1c) less than (<) 7 percentage (%) (Yes/No) | At week 104
  Measured as count of participants.
Participants acheiving body weight reduction greater than or equal to (>=) 5% (Yes/No) | At week 104
  Measured as count of participants.

SECONDARY OUTCOMES:
Change in HbA1c | From randomisation (week 0) to week 104
  Measured as percentage (%)-point.
Change in fasting plasma glucose (FPG) | From randomisation (week 0) to week 104
  Measured in millimoles per liter (mmol/l).
Change in self-measured plasma glucose (SPMG) 7-point mean profile | From randomisation (week 0) to week 104
  Measured in millimoles per liter(mmol/l).
Change in self-measured plasma glucose (SPMG) mean post prandial increments | From randomisation (week 0) to week 104
  Measured in millimoles per liter(mmol/l).
Time to additional anti-diabetic medication | From randomisation (week 0) to week 104
  Measured in days.
Change in body weight | From randomisation (week 0) to week 104
  Measured in kilograms (kg).
Relative change in body weight | From randomisation (week 0) to week 104
  Measured as percentage (%).
Change in waist circumference | From randomisation (week 0) to week 104
  Measured in centimeters (cm).
Participants achieving glycated haemoglobin (HbA1c) less than or equal to (<=) 6.5% (Yes/No) | From randomisation (week 0) to week 104
  Measured as count of participants.
Participants achieving glycated haemoglobin (HbA1c) reduction greater than or equal to (>=) 0.7%-point (Yes/No) | From randomisation (week 0) to week 104
  Measured as count of participants.
Participants achieving body weight reduction greater than or equal to (>=) 5 percentage (%) | From randomisation (week 0) to week 104
  Measured as count of participants.
Change in systolic blood pressure | From randomisation (week 0) to week 104
  Measured in millimiters of mercury (mmHg).
Change in total cholesterol | From randomisation (week 0) to week 104
  Measured as ratio to baseline.
Change in high density lipoprotein (HDL) | From randomisation (week 0) to week 104
  Measured as ratio to baseline.
Change in low density lipoprotein (LDL) | From randomisation (week 0) to week 104
  Measured as ratio to baseline.
Change in very low density lipoprotein (VLDL) | From randomisation (week 0) to week 104
  Measured as ratio to baseline.
Change in Triglycerides | From randomisation (week 0) to week 104
  Measured as ratio to baseline.
Change in free fatty acids | From randomisation (week 0) to week 104
  Measured as ratio to baseline.
Number of treatment emergent adverse events | From randomisation (week 0) to week 109
  Measured as count of events.
Change in Control of Eating Questionnaire (CoEQ) score - Craving Control domain | From randomisation (week 0) to week 104
  Measured as score on a scale. Scales range from 0 (minimum) to 10 (maximum).
Change in Control of Eating Questionnaire (CoEQ) score - Craving for Savory domaina | From randomisation (week 0) to week 104
  Measured as score on a scale. Scales range from 0 (minimum) to 10(maximum).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com